CLINICAL TRIAL: NCT06314906
Title: Combining Electroacupuncture With Antiemetic Therapy for Preventing Chemotherapy-Induced Nausea and Vomiting in Patients With Breast Cancer: A Clinical Study
Brief Title: Electroacupuncture Plus Antiemetic Therapy for Chemotherapy-Induced Nausea and Vomiting in Patients With Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Feixue Song (Other)
Responsible Party: Sponsor-Investigator, Feixue Song, Professor, Lanzhou University Second Hospital
Organization: Lanzhou University Second Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHLU-2024001
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Electroacupuncture; Olanzapine-contained Four-drug Antiemetic; Nausea and Vomiting
Keywords: electroacupuncture; olanzapine-contained four-drug antiemetic; nausea and Vomiting; breast cancer; chemotherapy
MeSH Terms: conditions — Nausea; Vomiting; Breast Neoplasms | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- True Acupuncture Combined with Antiemetic Therapy (Experimental): Participants in this arm will undergo electroacupuncture sessions once daily from day 1 to day 4. Electrical stimulation will be administered for 30 minutes at alternating frequencies of 2/10Hz.
  Interventions: Device: Electroacupuncture; Drug: Antiemetic Therapy
- Antiemetic therapy (Placebo Comparator): Participants assigned to this arm will receive sham electroacupuncture sessions daily from day 1 to day 4, mirroring the schedule of the experimental group. They will also receive the same antiemetic medications as the experimental group.
  Interventions: Device: Sham electroacupuncture; Drug: Antiemetic Therapy

INTERVENTIONS:
Device: Electroacupuncture — Participants in this arm will undergo electroacupuncture sessions once daily from day 1 to day 4. Electrical stimulation will be administered for 30 minutes at alternating frequencies of 2/10Hz
  Arms: True Acupuncture Combined with Antiemetic Therapy
Drug: Antiemetic Therapy — Participants will receive oral olanzapine at a dose of 5 mg per day on days 1 through 4, along with NK1 receptor antagonist, 5HT3 receptor antagonist, and intravenous dexamethasone at a dose of 10 mg 30 minutes prior to chemotherapy on Day 1, followed by intravenous dexamethasone at a dose of 8 mg on days 2, 3, and 4 post-chemotherapy.
  Arms: True Acupuncture Combined with Antiemetic Therapy
Device: Sham electroacupuncture — Participants assigned to this arm will receive sham electroacupuncture sessions daily from day 1 to day 4, mirroring the schedule of the experimental group
  Arms: Antiemetic therapy
Drug: Antiemetic Therapy — They will also receive the same antiemetic medications as the experimental group.
  Arms: Antiemetic therapy

SUMMARY:
This study explores the effectiveness of combining electroacupuncture with olanzapine-containing four-drug antiemetic therapy to mitigate chemotherapy-induced nausea and vomiting (CINV) in patients with breast cancer. The research aims to assess the adjunctive benefits of electroacupuncture in enhancing the antiemetic effects of conventional medication, particularly in the context of highly emetogenic chemotherapy regimens. By investigating the synergistic potential of these modalities, the study seeks to provide insights into optimizing supportive care strategies for patients with breast cancer undergoing intensive chemotherapy treatment.

DETAILED DESCRIPTION:
This study is a randomized controlled trial conducted in parallel groups, with blinding implemented. It aims to assess the effectiveness of combining electroacupuncture with standard quadruple antiemetic drugs for patients with breast cancer undergoing HEC.

Both study arms will be administered Olanzapine, Neurokinin-1 receptor antagonists, serotonin receptor antagonists, and dexamethasone at the commencement of HEC on Day 1. Subsequently, participants will be randomly assigned to receive either electroacupuncture or sham acupuncture.

Participants will be responsible for recording all instances of nausea and vomiting, as well as documenting the use of rescue antiemetic medications.

The study will evaluate primary and secondary outcomes, as well as monitor adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 75 years, inclusive, from any nationality.
2. Patients diagnosed with early-stage breast cancer.
3. Eastern Cooperative Oncology Group performance status ranging from 0 to 2.
4. All patients must undergo highly emetogenic chemotherapy (HEC).
5. Adequate organ function.
6. Adequate contraception required for premenopausal women.

Exclusion Criteria:

1. Scheduled to undergo chemotherapy between days 2 to 4 following HEC.
2. Received or is planned to receive abdominal radiation therapy within 1 week before Day 1 in cycle 1.
3. Significant medical or psychological conditions.
4. Presents with symptomatic primary or metastatic central nervous system malignancy causing nausea and/or vomiting.
5. Experiencing ongoing vomiting or nausea of grade 2 or higher according to Common Terminology Criteria for Adverse Events (CTCAE).
6. Any known allergies to the study drug, antiemetics, or dexamethasone.
7. Patients who have fear of electroacupuncture stimulation or are allergic to stainless steel needles.
8. Received acupuncture treatments for any conditions within 8 weeks prior to HEC.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients Free from Nausea Throughout Treatment | 120 hours
  The proportion of patients experiencing no nausea is determined by those who register a score of 0 on the visual-analogue scale for nausea throughout the entirety of treatment, spanning from initiation of chemotherapy to 120 hours post-treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Hospital of Lanzhou University, Lanzhou, Gansu, China